CLINICAL TRIAL: NCT06005792
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending-Dose Study of the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of XmAb27564 in Patients With Plaque Psoriasis and Atopic Dermatitis
Brief Title: Multiple Ascending-Dose Study of XmAb®27564 in Patients With Psoriasis or Atopic Dermatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XmAb27564-02
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis; Atopic Dermatitis
Keywords: Psoriasis; Plaque Psoriasis; Atopic Dermatitis; Eczema
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Plaque Psoriasis (Experimental)
  Interventions: Biological: XmAb27564; Biological: Placebo
- Atopic Dermatitis (Experimental)
  Interventions: Biological: XmAb27564; Biological: Placebo

INTERVENTIONS:
Biological: XmAb27564 — Subjects to receive four doses of XmAb27564 at one of six escalating dose-levels administered subcutaneously every 2 weeks (Q2W).
Biological: Placebo — Subjects to receive four doses of placebo administered subcutaneously every 2 weeks (Q2W).

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of XmAb27564 following multiple doses among participants with plaque psoriasis and atopic dermatitis.

DETAILED DESCRIPTION:
This is a phase 1b, randomized, double-blind, placebo-controlled, multiple ascending dose (MAD) study of XmAb27564. It is planned to enroll approximately 48 adult patients with mild-to-severe plaque psoriasis and 80 adult patients with moderate-to-severe atopic dermatitis. All patients will receive a total of 4 doses of study drug or placebo, administered subcutaneously every 2 weeks. A one year, open-label extension is available to qualifying patients.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion and exclusion criteria include, but are not limited to, the following:

* Have active mild-to-severe plaque psoriasis or moderate-to-severe atopic dermatitis according to study-specific criteria
* Weight between 40 to 150 kg, inclusive
* No topical treatments for psoriasis or atopic dermatitis for 2 weeks before randomization
* No phototherapy for psoriasis for 4 weeks before randomization
* Washout of oral treatments for psoriasis or atopic dermatitis for 4 weeks before randomization
* Washout of biologic treatments for psoriasis or atopic dermatitis for 12 weeks before randomization
* Stated willingness to comply with all study procedures (including skin biopsies) and availability for the duration of the study

Exclusion Criteria:

* Patients with a history of active asthma within 5 years of screening, except those that have well controlled asthma symptoms at screening visit.
* Patients who have had any prior investigational treatment with IL-2 therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple ascending dose subcutaneous (SC ) administration of XmAb27564 | Day 57
  Safety and tolerability will be assessed by incidence of AE's; incidence of clinically significant changes in physical exams, vital signs, ECGs, and clinical laboratory testing; incidence of DLT's

SECONDARY OUTCOMES:
To characterize pharmacokinetics | Day 57
  Pharmacokinetics will be assessed by serum XmAb27564 concentrations
To characterize pharmacodynamics | Day 57
  Pharmacodynamics will be assessed by the change in number of regulatory T cells, conventional T cells, and natural killer cells (NK cells) in blood

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Zitnik, MD, Study Director — Executive Medical Director, Clinical Development, Xencor, Inc.
Locations (7):
- United States (6):
  - Unison Clinical Trials, Sherman Oaks, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - Driven Research, Coral Gables, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - J&S Studies, Inc, College Station, Texas
  - Center for Clinical Studies, LTD. LLP, Webster, Texas
- Innovaderm Research Inc., Montreal, Quebec, Canada